CLINICAL TRIAL: NCT05134506
Title: Effects of a Structured Dance Program in Parkinson's Disease. A Greek Pilot Study
Brief Title: Dance in Parkinson's Disease. A Greek Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of West Attica (Other)
Responsible Party: Principal Investigator, Michail Elpidoforou, Principal Investigator, University of West Attica
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 296/24.4.2019
Record Dates: First submitted 2021-10-16; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Dance; Dance for Parkinson's; Quality of Life; Depression; Fatigue; Cognitive Functions
MeSH Terms: conditions — Parkinson Disease; Depression; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dance for PD® classes (Experimental): Dance for PD® was developed by the Brooklyn Parkinson Group (BPG) in collaboration with the Mark Morris Dance Group (MMDG) in 2001. It was designed to introduce people with PD to techniques used by dancers to control movement and it integrates different dance genres while participants dance individually and in groups rather than partnered.
  Interventions: Behavioral: Dance for PD® classes

INTERVENTIONS:
Behavioral: Dance for PD® classes — The intervention consisted of 16 60-min classes, performed twice weekly over a period of 8 weeks and instructed by a single researcher who had the approval to use it for research reasons.

SUMMARY:
Dance for Parkinson's Disease® (DfPD®) is a structured dance program that has never been evaluated in Greek PD population. This study assesses for the first time the efficacy, safety and feasibility of DfPD® program in Greek PD patients.

A total of 16 early-to-mid-stage PD patients underwent a total of 16 60-min classes of adjusted to Greek music and dance culture DfPD®, twice weekly, over 8 weeks. Assessments were performed at baseline and at the end of the study period and included quality of life, depressive symptoms, fatigue, cognitive functions, balance and body mass index. Safety and feasibility were also assessed.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is an idiopathic, neurodegenerative, and progressive movement disorder caused mainly by dysfunction of dopaminergic cells of the substantia nigra. Numerous studies demonstrate the benefits of regular physical exercise in PD, with aerobic exercise having a greater neuroprotective effect by stimulating brain neuroplasticity. People with PD are more easily motivated to attend dance classes systematically than other forms of exercise, they have a high compliance rate with low dropouts, and often continue to practice dance outside the dance intervention.

DfPD® (Dance for Parkinson's Disease®, or Dance for PD®) was developed by the Brooklyn Parkinson Group (BPG) in collaboration with the Mark Morris Dance Group (MMDG) in 2001.This intervention has previously been shown to exert beneficial effect on QoL, motor functions, cognition, self-efficacy, anxiety and depression in people with PD. To the investigators' knowledge, there is no study investigating the effect of any structured dance program in Greek PD patients. Furthermore, no study to date has investigated the effect of DfPD® on PD patients' fatigue. The present pilot study aimed at evaluating for the first time the efficacy, safety and feasibility of a culturally adjusted DfPD® program in Greek patients with early-to-mid-stage PD.

This is a prospective, non-randomized, uncontrolled, open-label, pilot study. A total of 16 early-to-mid-stage PD patients underwent a total of 16 60-min classes of adjusted to Greek music and dance culture DfPD®, twice weekly, over 8 weeks. Assessments were performed at baseline and at the end of the study period and included quality of life, depressive symptoms, fatigue, cognitive functions, balance and body mass index. Safety and feasibility were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* An established diagnosis of idiopathic PD of an early-to-moderate severity; that is from 0 to 2,5 according to Hoehn and Yahr (H&Y) stages
* Ability to understand, write and speak in Greek
* Written consent for participating into the study

Exclusion Criteria:

* A diagnosis of a non-PD tremor disorder
* Moderate-to-severe PD (≥3 H&Y stages) due to a high falls risk
* Serious health or disability issues (either physical or mental) due of which exercise is not permitted and/or basic instructions during the program cannot be followed
* Mental disorder not related to PD
* Any disease other than PD which could affect mobility levels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Change in total score of Parkinson's Disease Questionnaire-8 | Baseline (week 1), end of intervention (week 10)
  Minimum score 0, Maximum score 100. A higher score indicates worse quality of life.
Occurence of Emergent Adverse Events | During the intervention (week 2-9)
  Occurrence of adverse events comprising falls, injuries, muscle soreness or excessive fatigue.
Financial Feasibility Assessment | During the intervention (week 2-9)
  No cost for the studio and the dance instructor.
Adherence and Attrition Assessment | During the intervention (week 2-9)
  Adherence and attrition rates; an adherence rate ≥70% is considered as high in elderly with functional limitations, and attrition rate ≤15% is considered acceptable by the PEDro scale.
Assessment of Willingness to Continue the Program after the Intervention | End of intervention (week 10)
  Verbal statement for continuing the program after the end of the intervention
Assessment of Recruitment Rates | Start of Recruitment (-3 months), Baseline (week 1)
  Target, up to 2 months for 16 participants.

SECONDARY OUTCOMES:
Change in total score of Beck Depression Inventory-II | Baseline (week 1), end of intervention (week 10)
  Minimum score 0, Maximum score 63. A higher score indicates worse depressive symptoms.
Change in total score of Parkinson Fatigue Scale-16 | Baseline (week 1), end of intervention (week 10)
  Minimum score 1, Maximum score 5. A higher score indicates more fatigue.
Change in total score of Montreal Cognitive Assessment | Baseline (week 1), end of intervention (week 10)
  Minimum score is 0, Maximum score 30. Lower scores indicate cognitive impairment.
Change in total score of Berg Balance Scale | Baseline (week 1), end of intervention (week 10)
  Minimum score is 0, Maximum score is 56. Lower scores indicate worse balance.
Change in Body Mass Index | Baseline (week 1), end of intervention (week 10)
  Lower scores than 18,5 indicate underweight, scores of 18,5-24,9 indicate normal weight, scores of 25-29,9 indicate overweight and scores of over 30 indicate obesity.

CONTACTS AND LOCATIONS:
Overall Officials: Michail Elpidoforou, MSc, Principal Investigator — Laboratory of Neuromuscular and Cardiovascular Study of Motion (LANECASM)
Locations (1):
- Laboratory of Neuromuscular and Cardiovascular Study of Motion (LANECASM), Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No